CLINICAL TRIAL: NCT03447470
Title: A Modular Multi-Arm, Phase 1, Adaptive Design Study to Evaluate the Safety and Tolerability of RXC004, Alone and in Combination With Anti-cancer Treatments, in Patients With Advanced Malignancies
Brief Title: Study to Evaluate the Safety and Tolerability of RXC004 in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Redx Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RXC004/0001
Record Dates: First submitted 2018-02-14; First posted 2018-02-27 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Solid Tumor
Keywords: Biliary tract cancers; Thymus cancers
MeSH Terms: conditions — Neoplasms; Biliary Tract Neoplasms; Thymus Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Module 1 monotherapy Dose escalation in those patients with advanced solid tumors while being monitored for safety and dose-limiting toxicity. This module will provide information on dosing and schedules for further module(s).
  Module 2 will commence by enrolling patients with advanced solid tumors into a monotherapy dose escalation, in combination with a fixed dose of nivolumab (a known anti-cancer treatment). This module will provide information and safety and tolerability of the study drug or in combination with the anti-cancer treatment.
  Module 3 will investigate the pharmacokinetic, Wnt pathway inhibition, incidence/severity of Wnt pathway related adverse events and anti-tumour activity of RXC004 when given at 2 different intermittent dosing schedules in selected patients with Wnt ligand dependent advanced tumours.
Masking Description: Open label design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg) (Experimental): Patients were given 0.5 mg RXC004 and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004
- Module 2 Arm 1 - RXC004 (1.0 mg) plus Nivolumab (Experimental): Patients were given 1.0 mg RXC004 in combination with a standard dose of Nivolumab and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004; Drug: Nivolumab
- Module 3 - Intermittent schedules of monotherapy RXC004 (Experimental): Patients were given 2.0 mg RXC004. The patients were treated for 2 weeks at the same dose, followed by 1 week off for a 21 day cycle.
  Interventions: Drug: RXC004
- Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg) (Experimental): Patients were given 1.0 mg RXC004 and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004
- Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg) (Experimental): Patients were given 1.5 mg RXC004 and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004
- Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg) (Experimental): Patients were given 2.0 mg RXC004 and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004
- Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg) (Experimental): Patients were given 3.0 mg RXC004 and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004
- Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg) (Experimental): Patients were given 10.0 mg RXC004 and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004
- Module 2 Arm 2 - RXC004 (1.5 mg) plus Nivolumab (Experimental): Patients were given 1.5 mg RXC004 in combination with a standard dose of Nivolumab and monitored for Dose Limiting Toxicities.
  Interventions: Drug: RXC004; Drug: Nivolumab

INTERVENTIONS:
Drug: RXC004 — RXC004 is taken orally, inhibits porcupine (PORCN) and interacts with the wnt signalling pathway.
Drug: Nivolumab — RXC004 is taken orally, inhibits porcupine (PORCN) and interacts with the wnt signalling pathway.
  Nivolumab is a fully human monoclonal immunoglobulin G4 antibody to PD-1
  Arms: Module 2 Arm 1 - RXC004 (1.0 mg) plus Nivolumab; Module 2 Arm 2 - RXC004 (1.5 mg) plus Nivolumab

SUMMARY:
The purpose of this study is to determine the safety and tolerability of RXC004 as monotherapy and in combination with Nivolumab in patients with advanced malignancies. In order to define the doses and schedules for further clinical evaluation.

DETAILED DESCRIPTION:
The study will consist of an ascending monotherapy dose, the doses are pre-defined.

The decision to escalate will be made upon the assessment of safety and tolerability data in the first cycle of treatment.

Module 1 will commence with a 3+3 dose escalation design up to a recommended Phase 2 monotherapy dose. Patients being monitored for dose limiting toxicities at each dose level.

Characterisation of the PK profile, MTD and/or recommended Phase 2 dose will be defined on the emerging data.

Module 2: RXC004 and Nivolumab - Follows a similar 3+3 dose escalation design using RXC004 plus Nivolumab. The MTD and/or Phase 2 dose will be defined based on the PK profile, emerging safety and the appearance of any dose limiting toxicities.

Module 3: Intermittent dose schedules of RXC004 will be investigated. The intermittent schedules will utilize the module 1 dose which was shown to be safe and tolerated when used continuously. Characterisation of the PK profile; Wnt pathway inhibition; incidence/severity of Wnt pathway related AEs and anti-tumor activity will be evaluated at 2 different dosing schedules.

ELIGIBILITY:
(Summarized due to limitation of characters)

Inclusion Criteria:

* Written informed consent
* Aged at least 18 years
* Histological or cytological confirmation of advanced malignancy not considered to be appropriate for further conventional treatment
* Patients must use adequate contraception measures for the duration of the study and for 6 months after the study
* Patients must have adequate organ functions
* Ability to swallow and retain oral medication

Exclusion Criteria:

* Prior treatment with a compound of the same mechanism of action as RXC004
* No other anti-cancer therapy or investigational product throughout the study
* Patients with persistent grade 2 or higher diarrhoea
* Patients at high risk of bone fractures
* QTc prolongation
* Known uncontrolled intercurrent illness
* Known severe allergies to any active or inactive ingredients

In addition for Module 2

* Patients with any contraindication/hypersensitivity to Nivolumab of excipients
* Patients with active or prior documented autoimmune of inflammatory disorders within the past 5 years
* Patients with active infections, including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus
* Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of initiation of study treatment
* Patients with body weight <40kg
* Patients with a history of allogeneic organ transplant or active primary immunodeficiency

In addition to Module 3

Patients with Wnt ligand-dependent solid tumours, defined as:

* Biliary tract cancers
* Thymus cancers (thymic and thymoma WHO classification)
* Any solid tumour with documented aberration in RNF43 and/or RSPO from central pre-screening or from a recognised panel approved by the Sponsor
* Patients willing to have mandatory skin biopsies at baseline and on one occasion while on study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Cook, Principal Investigator — The Christie NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Royal Marsden Hospital, Institute of Cancer Research, Sutton, Surrey
  - Guys Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle
  - Department of Oncology, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into one of the modules of the study.
Pre-assignment Details: In Module 1, participants enrolled, into 6 arms at different dose levels: 0.5 mg; 1 mg; 1.5 mg; 2 mg; 3 mg; 10 mg.
  In Module 2, participants enrolled, into 2 arms at different dose levels (1.0 mg and 1.5 mg) of RXC004 in combination with Nivolumab.
  In Module 3, the enrolled participants received a dose of 2.0 mg of RXC004 at 2 weeks on/1 week off.
Groups:
- Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg): Patients were given 0.5 mg RXC004 monitored for Dose Limiting Toxicities.
- Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg): Patients were given 1.0 mg RXC004 monitored for Dose Limiting Toxicities.
- Module 3 - Intermittent Schedules of Monotherapy RXC004: Patients were given RXC004 at 2 mg once a day (QD) for 2 weeks, followed by 1 week off for 21 day treatment cycles.
Period: Overall Study
Arm/Group | Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg) | Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg) | Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg) | Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg) | Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg) | Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg) | Module 2 Arm 1 - RXC004 (1.0 mg) Plus Nivolumab | Module 2 Arm 2 - RXC004 (1.5 mg) Plus Nivolumab | Module 3 - Intermittent Schedules of Monotherapy RXC004
Started | 4 | 3 | 7 | 6 | 4 | 1 | 6 | 8 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 7 | 6 | 4 | 1 | 6 | 8 | 7
Not completed — Death | 0 | 1 | 3 | 0 | 1 | 0 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Not completed — Treatment discontinued | 3 | 2 | 4 | 6 | 2 | 1 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population described here per module include: In Module 1, participants enrolled, into 6 arms at different dose levels: 0.5 mg; 1 mg; 1.5 mg; 2 mg; 3 mg; 10 mg.
  In Module 2, participants enrolled, into 2 arms at different dose levels (1.0 mg and 1.5 mg) of RXC004 in combination with Nivolumab.
  In Module 3, the enrolled participants received a dose of 2.0 mg of RXC004 at 2 weeks on/1 week off.
Groups:
- Intermittent Schedules of Monotherapy RXC004 - Module 3: Patients were given RXC004 at 2 mg once a day (QD). Patients were treated for 2 weeks at the same dose, followed by 1 week off for 21 day treatment cycles.
- Total: Total of all reporting groups
Arm/Group | Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg) | Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg) | Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg) | Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg) | Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg) | Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg) | Module 2 Arm 1 - RXC004 (1.0 mg) Plus Nivolumab | Module 2 Arm 2 - RXC004 (1.5 mg) Plus Nivolumab | Intermittent Schedules of Monotherapy RXC004 - Module 3 | Total
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 4 | 1 | 6 | 8 | 7 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4 | 2 | 1 | 1 | 4 | 4 | 4 | 24
  >=65 years | 3 | 0 | 3 | 4 | 3 | 0 | 2 | 4 | 3 | 22
Age, Continuous [Median (Full Range); unit: Years] | 73 [60 to 76] | 57 [44 to 62] | 62 [46 to 77] | 67 [56 to 73] | 68.5 [60 to 75] | 59 [59 to 59] | 46.5 [39 to 74] | 64.5 [30 to 75] | 63 [42 to 84] | 63.2 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 2 | 3 | 0 | 5 | 2 | 4 | 22
  Male | 2 | 2 | 4 | 4 | 1 | 1 | 1 | 6 | 3 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 3
  White | 4 | 3 | 6 | 4 | 3 | 1 | 5 | 7 | 7 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Module 1 - Safety and Tolerability of RXC004 by Assessment of Whether Any Dose Limiting Toxicities (DLT) Arise From First Dose Until the End of 21 Days of Continuous Dosing:
Description: A DLT was defined as an adverse event or abnormal laboratory value. Haematological toxicity of CTCAE grade 4 or higher for more than 4 consecutive days.
  Grade 3 neutropenia of any duration accompanied by fever 38.5 degrees Celsius or higher.
  Grade 3 thrombocytopaenia with bleeding. Any other confirmed haematological toxicity CTCAE grade 4 or higher. Non-haematological toxicity CTCAE grade 3 or higher. Any other toxicity that is judged to be a DLT by the Safety Review Committee. An AE resulting in disrupted dosing >14 days.
Time Frame: AE data was collected after each cycle and until 30-day follow-up visit after study exit. The DLT period were assessed from the first dose until the end of 21 days of continuous dosing in each cycle until a Maximum Tolerated Dose (MTD) was identified.
Population: RXC004 monotherapy was evaluated at 6 increasing doses.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg) | Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg) | Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg) | Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg) | Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg) | Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 4 | 1
Participants
  Patients with any DLT | 0 | 0 | 0 | 1 | 2 | 1
  Colitis | 0 | 0 | 0 | 0 | 1 | 0
  Diarrhoea | 0 | 0 | 0 | 0 | 0 | 1
  Enteritis | 0 | 0 | 0 | 0 | 1 | 0
  Pancreatitis | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Module 2 - Safety and Tolerability of RXC004 in Combination With Nivolumab by Assessment of Whether Any Dose Limiting Toxicities (DLT) Arise From First Dose Until the End of 28 Days of Continuous Dosing.
Description: A DLT is defined as an adverse event or abnormal laboratory value. Haematological toxicity of CTCAE grade 4 or higher for more than 4 consecutive days.
  Grade 3 neutropenia of any duration accompanied by fever 38.5 degrees Celsius or higher.
  Grade 3 thrombocytopaenia with bleeding. Any other confirmed haematological toxicity CTCAE grade 4 or higher. Non-haematological toxicity CTCAE grade 3 or higher. Any other toxicity that is judged to be a DLT by the Safety Review Committee. An AE resulting in disrupted dosing >14 days. Any grade 3 or higher immune-related adverse events
Time Frame: The DLT period will be assessed from the first dose until the end of 28 days of continuous dosing. This will be completed for each dose level until a Maximum Tolerated Dose (MTD) is identified. Estimated time 12 Months in total
Population: RXC004 (at 2 doses) was evaluated in combination with Nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 2 Arm 1 - RXC004 (1.0 mg) Plus Nivolumab | Module 2 Arm 2 - RXC004 (1.5 mg) Plus Nivolumab
Number analyzed (Participants) | 5 | 6
Participants
  Patients with any DLT | 0 | 1
  Drug-induced Liver Injury | 0 | 1

3. Primary Outcome: Module 3 - Safety and Tolerability of RXC004 at Intermittent Dosing Schedule.
Description: Haematological toxicity of CTCAE grade 4 or higher present for more than 4 consecutive days.
  Grade 3 neutropenia of any duration accompanied by fever 38.5 degrees Celsius or higher.
  Grade 3 thrombocytopaenia with bleeding. Any other confirmed haematological toxicity CTCAE grade 4 or higher. Non-haematological toxicity CTCAE grade 3 or higher. Any other toxicity that is judged to be a DLT by the Safety Review Committee. An AE resulting in disrupted dosing >14 days. Any grade 3 or higher immune-related adverse events.
Time Frame: The assessment period will be from the first dose until the end of 21 days of intermittent dosing or within 7 days of IP discontinuation.
Population: RXC004 was evaluated at a dose of 2 mg monotherapy administered as an intermittent schedule of 2 weeks on/1 week off dosing
Measure: Count of Participants; unit: Participants
Arm/Group | Module 3 - Intermittent Schedules of Monotherapy RXC004
Number analyzed (Participants) | 7
Participants | 0

4. Secondary Outcome: Module 1 - PK Profile - AUC on Cycle 0 Day 1 (C0D1)
Description: Area under the Curve, AUC (0-24) for RXC004 was calculated from the measurement of mean plasma concentration of RXC004 at various time points from 0 - 96 hours following single dose on Cycle 0 Day1.
Time Frame: Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter AUC (0-24) was analyzed at various dose levels ranging from 0.5 - 10 mg.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Groups:
- Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg): Patients were given 0.5 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg): Patients were given 1.0 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg): Patients were given 1.5 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg): Patients were given 2.0 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg): Patients were given 3.0 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg): Patients were given 10 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
Arm/Group | Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg) | Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg) | Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg) | Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg) | Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg) | Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg)
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 4 | 1
h*ng/ml | 138.8 (27.9) | 334.8 (118.8) | 464.9 (223.2) | 552.5 (215.3) | 1350.6 (217.8) | 2702.2

5. Secondary Outcome: Module 1 - PK Profile - C24 on Cycle 0 Day 1 (C0D1)
Description: Mean Plasma concentration of RXC004 at 24 h post-dose calculated from the measurement of mean RXC004 concentrations at various time points from 0 - 96 hours following single dose on Cycle 0 Day1..
Time Frame: Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter, C24, was analyzed at various dose levels ranging from 0.5 - 10 mg.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- 0.5 mg: Patients were given 0.5 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- 1 mg: Patients were given 1.0 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- 1.5 mg: Patients were given 1.5 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- 2 mg: Patients were given 2.0 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- 3 mg: Patients were given 3.0 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
- 10 mg: Patients were given 10 mg RXC004. Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters.
Arm/Group | 0.5 mg | 1 mg | 1.5 mg | 2 mg | 3 mg | 10 mg
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 4 | 1
ng/ml | 1.74 (0.86) | 5.28 (3.66) | 7.26 (4.67) | 6.55 (4.62) | 16.05 (4.71) | 49.5

6. Secondary Outcome: Module 1 - PK Profile - Cmax on Cycle 0 Day 1 (C0D1)
Description: Maximum plasma concentration (Cmax) of RXC004 following single dose calculated from the measurement of mean plasma concentration of RXC004 at various time points from 0 - 96 hours following single dose on Cycle 0 Day1..
Time Frame: Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter Cmax was analyzed at various dose levels ranging from 0.5 - 10 mg.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 0.5 mg | 1 mg | 1.5 mg | 2 mg | 3 mg | 10 mg
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 4 | 1
ng/ml | 20.58 (3.07) | 47.77 (18.68) | 69.59 (33.1) | 84.03 (36.83) | 198.50 (57.81) | 369

7. Secondary Outcome: Module 1 - PK Profile - Half-life From PK Analysis on Cycle 0 Day 1 (C0D1)
Description: Half-life of RXC004 following single dose on Cycle 0 Day1 calculated from the measurement of mean plasma concentration of RXC004 at various time points from 0 - 96 hours following single dose on Cycle 0 Day1..
Time Frame: Samples were analyzed from 0 - 96 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter Half-life was analyzed at various dose levels ranging from 0.5 - 10 mg.
Measure: Median (Full Range); unit: hours
Arm/Group | 0.5 mg | 1 mg | 1.5 mg | 2 mg | 3 mg | 10 mg
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 4 | 1
hours | 16.77 [11.8 to 30.2] | 15.04 [8.5 to 21.2] | 16.88 [7.8 to 22.5] | 15.37 [9.9 to 21.2] | 14.44 [11.6 to 26.3] | 20.0

8. Secondary Outcome: Module 2 - PK Profile - AUC on Cycle 0 Day 1 (C0D1)
Description: AUC was calculated from the measurement of mean plasma concentration of RXC004 at various time points from 0 - 48 hours following single dose of RXC004 in combination with Nivolumab on Cycle 0 Day1.
Time Frame: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter AUC(0-24) was analyzed at the indicated dose levels.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Groups:
- 1 mg + Nivolumab: Patients were given 1.0 mg RXC004 plus Nivolumab. Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters.
- 1.5 mg + Nivolumab: Patients were given 1.5 mg RXC004 plus Nivolumab. Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters.
Arm/Group | 1 mg + Nivolumab | 1.5 mg + Nivolumab
Number analyzed (Participants) | 6 | 8
h*ng/ml | 303.3 (93.57) | 431.23 (109.63)

9. Secondary Outcome: Module 2 - PK Profile - C24 on Cycle 0 Day 1 (C0D1)
Description: Mean Plasma concentration of RXC004 at 24 h post-dose when given in combination with Nivolumab.
Time Frame: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter C24 was analyzed at the indicated dose levels.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 1 mg + Nivolumab | 1.5 mg + Nivolumab
Number analyzed (Participants) | 6 | 8
ng/ml | 6.18 (6.75) | 7.54 (3.12)

10. Secondary Outcome: Module 2 - PK Profile - Cmax on Cycle 0 Day 1 (C0D1)
Description: Maximum plasma concentration (Cmax) of RXC004 following single dose on Cycle 0 Day1 when given in combination with Nivolumab..
Time Frame: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter Cmax was analyzed at the indicated dose levels.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 1 mg + Nivolumab | 1.5 mg + Nivolumab
Number analyzed (Participants) | 6 | 8
ng/ml | 49.63 (13.55) | 50.93 (18.15)

11. Secondary Outcome: Module 2 - PK Profile - Half-life From PK Analysis on Cycle 0 Day 1 (C0D1)
Description: Half-life of RXC004 following single dose on Cycle 0 Day1 when given in combination with Nivolumab.
Time Frame: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter Half-life was analyzed at the indicated dose levels.
Measure: Median (Full Range); unit: hours
Arm/Group | 1 mg + Nivolumab | 1.5 mg + Nivolumab
Number analyzed (Participants) | 5 | 7
hours | 16.35 [9.9 to 22.1] | 10.31 [7.1 to 14.5]

12. Secondary Outcome: Module 3 - PK Profile - AUC on Cycle 0 Day 1 (C0D1)
Description: AUC was calculated from the measurement of mean plasma concentration of RXC004 at various time points from 0 - 48 hours following single dose of RXC004
Time Frame: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter AUC (0-24) was analyzed at the indicated dose level.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Groups:
- 2.0 mg (2 Weeks on/1 Week Off Dosing): Patients were given RXC004 at 2 mg once a day (QD). Patients were treated for 2 weeks at the same dose, followed by 1 week off for 21 day treatment cycles.
  Samples were analyzed from 0-48 hours after administration to evaluate PK parameters.
  RXC004: RXC004 taken orally, inhibits porcupine (PORCN) and interacts with the wnt signaling pathway.
Arm/Group | 2.0 mg (2 Weeks on/1 Week Off Dosing)
Number analyzed (Participants) | 7
h*ng/ml | 547.51 (160.18)

13. Secondary Outcome: Module 3 - PK Profile - C24 on Cycle 0 Day 1 (C0D1)
Description: Mean Plasma concentration of RXC004 at 24 h post-dose
Time Frame: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter C24 was analyzed at the indicated dose level.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 2.0 mg (2 Weeks on/1 Week Off Dosing)
Number analyzed (Participants) | 7
ng/ml | 7.65 (3.6)

14. Secondary Outcome: Module 3 - PK Profile - Cmax on Cycle 0 Day 1 (C0D1)
Description: Maximum plasma concentration (Cmax) of RXC004 following single dose
Time Frame: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Population: PK parameter Cmax was analyzed at the indicated dose level.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 2.0 mg (2 Weeks on/1 Week Off Dosing)
Number analyzed (Participants) | 7
ng/ml | 84.87 (34.56)

15. Secondary Outcome: Module 3 - PK Profile - Half-life on Cycle 0 Day 1 (C0D1)
Description: Half-life of RXC004 following single dose.
Time Frame: Cycle 0 Day 1
Population: Samples were analyzed from 0 - 48 hours after administration to evaluate PK parameters on Cycle 0 Day 1.
Measure: Median (Full Range); unit: hours
Arm/Group | 2.0 mg (2 Weeks on/1 Week Off Dosing)
Number analyzed (Participants) | 7
hours | 10.5 [8.8 to 14.9]

ADVERSE EVENTS:
Time Frame: AE data was collected after each cycle and until 30-day follow-up visit after the last dose or study exit. The median duration of exposure for Module 1 was 7.0 weeks across all dose cohorts. For Module 2 - 7.1 weeks in the 1.0 mg group and 8.4 weeks in the 1.5 mg group; Module 3 - 5.0 weeks.
Groups:
- Intermittent Schedules of Monotherapy RXC004 - Module 3: Patients were given RXC004 at 2 mg once a day (QD). Patients were treated for 2 weeks at the same dose, followed by 1 week off for 21 day treatment cycles.
  RXC004: RXC004 taken orally, inhibits porcupine (PORCN) and interacts with the wnt signaling pathway.
Arm/Group | Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg) | Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg) | Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg) | Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg) | Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg) | Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg) | Module 2 Arm 1 - RXC004 (1.0 mg) Plus Nivolumab | Module 2 Arm 2 - RXC004 (1.5 mg) Plus Nivolumab | Intermittent Schedules of Monotherapy RXC004 - Module 3
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/3 | 3/7 | 0/6 | 1/4 | 0/1 | 3/6 | 3/8 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3 | 5/7 | 1/6 | 3/4 | 1/1 | 4/6 | 4/8 | 4/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/7 | 0/6 | 0/4 | 0/1 | 0/6 | 0/8 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1 Arm 1 - Monotherapy RXC004 (0.5 mg) (N=4) | Module 1 Arm 2 - Monotherapy RXC004 (1.0 mg) (N=3) | Module 1 Arm 3 - Monotherapy RXC004 (1.5 mg) (N=7) | Module 1 Arm 4 - Monotherapy RXC004 (2.0 mg) (N=6) | Module 1 Arm 5 - Monotherapy RXC004 (3.0 mg) (N=4) | Module 1 Arm 6 - Monotherapy RXC004 (10.0 mg) (N=1) | Module 2 Arm 1 - RXC004 (1.0 mg) Plus Nivolumab (N=6) | Module 2 Arm 2 - RXC004 (1.5 mg) Plus Nivolumab (N=8) | Intermittent Schedules of Monotherapy RXC004 - Module 3 (N=7)
Lung Infection/Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT03447470/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT03447470/SAP_001.pdf